CLINICAL TRIAL: NCT04368975
Title: Main Features and Ventilatory Management of Patients With ARDS Caused by COVID-19
Brief Title: ARDS Caused by COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Ubikare (Industry)
Responsible Party: Principal Investigator, Carlos Ferrando Ortolá, Head of Surgical Intensive Care Unit, Hospital Clinic of Barcelona
Other Study IDs: COVID-19 ARDS
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Acute Respiratory Failure With Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with the acute respiratory distress syndrome (ARDS) have markedly varied clinical presentations. Main characteristics of mechanically ventilated ARDS caused by COVID-19, and adherence to lung-protective ventilation strategies are not well known.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study in consecutive, mechanically ventilated patients with ARDS caused by COVID-19 (as defined by the Berlin criteria and confirmed COVID-19 infection in a respiratory tract sample), admitted into a network of 27 Spanish and Andorran intensive care units (ICUs). Clinical features, ventilatory management, and clinical outcomes will be examined

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* intubated and mechanically ventilated
* confirmed COVID-19 infection in a respiratory tract sample
* acute onset of ARDS, as defined by the Berlin criteria

Exclusion Criteria:

* patients with non-confirmed SARS-CoV-2 infection according to WHO guidance
* patients with no information on respiratory parameters
* non- intubated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with acute respiratory failure requiring invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Discontinuation from mechanical ventilation | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ferrando, Principal Investigator — Medical Research and Clinical Consulting
Locations (1):
- Ricard Mellado, Barcelona, Spain

REFERENCES:
- [Derived] Ferrando C, Suarez-Sipmann F, Mellado-Artigas R, Hernandez M, Gea A, Arruti E, Aldecoa C, Martinez-Palli G, Martinez-Gonzalez MA, Slutsky AS, Villar J; COVID-19 Spanish ICU Network. Clinical features, ventilatory management, and outcome of ARDS caused by COVID-19 are similar to other causes of ARDS. Intensive Care Med. 2020 Dec;46(12):2200-2211. doi: 10.1007/s00134-020-06192-2. Epub 2020 Jul 29. PMID 32728965